CLINICAL TRIAL: NCT00856921
Title: To Find Out the Genetic Relationship Between the Early-Onset Achalasia and AAAS Gene
Brief Title: Genetic Evaluation of AAAS Gene in Early-Onset Achalasia and Alacrima Patients
Acronym: AAAS
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Kee Wook Jung, Asan Medical Center
Other Study IDs: AAASachalasia
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Achalasia; Alacrima
Keywords: Relationship between achalasia and AAAS gene
MeSH Terms: conditions — Esophageal Achalasia; Alacrima

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA and genetic analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The AAAS gene has been known to cause achalasia, alacrima, adrenal abnormalities and a progressive neurological syndrome. A considerable proportion of achalasia patients have been known to show alacrima (decreased secretion of tears). However, the genetic mechanism between achalasia and alacrima has not been defined yet. The investigators postulated that some proportions of early-onset achalasia could be correlated with AAAS gene; thus, the investigators aimed to investigate the relationship between the AAAS gene and early-onset achalasia.

ELIGIBILITY:
Inclusion Criteria:

* early age onset
* primary achalasia patient
* less than 35 years old

Exclusion Criteria:

* secondary achalasia patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Early age onset achalasia
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Genetic relationship between achalasia and AAAS gene